CLINICAL TRIAL: NCT03608059
Title: Shanghai General Hospital Affiliated to Shanghai Jiao Tong University
Brief Title: ATG/PTCy in Haplo-PBSCT Randomized Controlled,Multi-center
Acronym: ATG/PTCy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SHSYXY-ATG/PTCy multi-center
Record Dates: First submitted 2018-07-28; First posted 2018-07-31 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Myeloid Tumor
Keywords: ATG; PTCy; haplo-PBSCT; GVHD

STUDY DESIGN:
Intervention Model Description: ATG+PTCy
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ATG/PTCy (Experimental): The GvHD prophylaxis consisted of ATG 2.5mg/kg administered on day -2 to -1 and cyclophosphamide (Cy) 50 mg/kg on day +3, cyclosporine A (CsA) and mycophenolate mofetil (MMF) initiating on day +4. CsA was prescribed at 2 mg/kg as a continuous infusion. The CsA doses were modified to obtain nadir serum levels between 200 and 300 ng/ml. MMF was administered at 15 mg/kg oral 3 times per day (maximum dose 3g per day) until day +34 and was then stopped if no aGvHD. Mycophenolate Sodium Enteric-coated Tablets (MPA) can be used instead of MMF, one tablet MPA corresponds to one tablet MMF. CsA was tapered from day +90 to day +180.
  Interventions: Drug: ATG/PTCy
- standard ATG (Active Comparator): The GvHD prophylaxis consisted of ATG 2.5mg/kg administered on day -4 to -1 , cyclosporine A (CsA) initiating on day -5 and mycophenolate mofetil (MMF) initiating on day +1 . CsA was prescribed at 2 mg/kg as a continuous infusion. The CsA doses were modified to obtain nadir serum levels between 200 and 300 ng/ml. MMF was administered at 15 mg/kg oral 2 times per day (maximum dose 2g per day) until day +30 and was then stopped if no aGvHD. Mycophenolate Sodium Enteric-coated Tablets (MPA) can be used instead of MMF, one tablet MPA corresponds to one tablet MMF. CsA was tapered from day +90 to day +180.
  Interventions: Drug: standard ATG
- standard PTCy (Active Comparator): The GvHD prophylaxis consisted of cyclophosphamide (Cy) 50 mg/kg on day +3, +4,cyclosporine A (CsA) and mycophenolate mofetil (MMF) initiating on day +5. CsA was prescribed at 2 mg/kg as a continuous infusion. The CsA doses were modified to obtain nadir serum levels between 200 and 300 ng/ml. MMF was administered at 15 mg/kg oral 3 times per day (maximum dose 3g per day) until day +35 and was then stopped if no aGvHD. Mycophenolate Sodium Enteric-coated Tablets (MPA) can be used instead of MMF, one tablet MPA corresponds to one tablet MMF. CsA was tapered from day +90 to day +180.
  Interventions: Drug: standard PTCy

INTERVENTIONS:
Drug: ATG/PTCy — low dose Antithymocyte Globulin plus low dose post-transplant cyclophosphamide as graft-versus-host disease prophylaxis in haploidentical peripheral blood stem cell transplantation
  Arms: ATG/PTCy
Drug: standard ATG — in vivo T cell depletion (TCD) with anti-thymocyte globulin (ATG) as graft-versus-host disease prophylaxis in haploidentical peripheral blood stem cell transplantation
  Other Names: ATG
  Arms: standard ATG
Drug: standard PTCy — post-transplant cyclophosphamide (PTCy) as graft-versus-host disease prophylaxis in haploidentical peripheral blood stem cell
  Other Names: PTCy
  Arms: standard PTCy

SUMMARY:
A novel regimen, which is composed of a low dose of ATG (5 mg/kg) and low-dose PTCy (one dose of PTCy, 50mg/kg) for GvHD prophylaxis in Haplo-PBSCT for patients with hematologic malignancies, was designed to decrease the risk of aGvHD and lower the incidence of virus reactivation.

DETAILED DESCRIPTION:
Acute graft-versus-host disease (aGvHD) is the most important obstacle of haploidentical hematopoietic stem cell transplantation (Haplo-HSCT) for treatment of patients with hematologic malignancies. In the last two decades, the results of Haplo-HSCT have been conspicuously improved due to effective prophylaxis strategies for aGvHD, such as in vivo T cell depletion (TCD) with anti-thymocyte globulin (ATG) or post-transplant cyclophosphamide (PTCy).

The regimens for prophylaxis of GvHD based on rabbit anti-human thymocyte immunoglobin (ATG 10mg/kg, Thymoglobin®, Genzyme Polyclonals S.A.S) effectively prevented the occurrence of grade II-IV aGvHD with an incidence of 33.4%-46%, grade III-IV aGvHD 12%-14.9%, but the reactivation incidences of cytomegalovirus (CMV) and EB virus (EBV) were higher due to a slower immune reconstitution(2-4). The 100-day CIs of CMV and EBV viremia were 61%-64%and over 50%, respectively. Although ATG-based regimens have achieved excellent results, the incidences of aGvHD and the post-transplant virus reactivation are still higher, affecting the long-term survival of the patients.

The regimen of PTCy for prevention of GvHD was developed in 1999 by St. Johns Hopkin's group in Baltimore (1) and had outstanding results with the CIs of 34% grades II-IV and of 6% grades III-IV aGvHD by day 200 in haplo-bone marrow transplantation (Haplo-BMT) (7), respectively. The incidences of viral and fungal infection in Haplo-HSCT with PTCy for GvHD prophylaxis were much lower than ATG based regimens. Ruggeri A（8）et al retrospectively analyzed the effects of different stem cell source (BM vs PBSC) on the transplant results in Haplo-HSCT with PTCy. The results showed that BM was associated with a lower incidence of grades II-IV and grades III-IV acute GVHD (21% vs 38%, P ≤ .01; and 4% vs 14%, P < .01, respectively), which was further confirmed by Bashey A et al' study（9）. These data indicated that PTCy regimen don't have the same effects for GvHD prophylaxis with PBSC graft as compared with BM graft in Haplo-HSCT.

A novel regimen, which is composed of a low dose of ATG (5 mg/kg) and low-dose PTCy (one dose of PTCy, 50mg/kg) for GvHD prophylaxis in Haplo-PBSCT for patients with hematologic malignancies, was designed to decrease the risk of aGvHD and lower the incidence of virus reactivation. A prospective, phase II clinical trial (Clinicaltrials.org NCT03395860) was performed to evaluate the efficacy with low dose ATG followed by low dose PTCy as GvHD prophylaxis.Thirty-two patients diagnosed with hematological malignancies were enrolled in this trial. All patients received myeloablative conditioning regimens except for three patients. The cumulative incidences (CIs) of grades II-IV and III-IV acute GvHD were 19.4% (95% CI, 5.5-33.3%) and 6.9% (95% CI 0-16.3%) by day 100, respectively. The one-year probability of relapse was 25.1% (95% CI, 7.3-42.9%). The one-year probabilities of disease free-survival (DFS) and overall survival (OS) was 59% (95% CI, 33.3%-84.7%) and 78.4% (95% CI, 63%-93.8%), respectively. The CIs of CMV reactivation and EBV reactivation by day 180 were 37.5% (95% CI, 19.8-55.2%) and 40.6% (95% CI, 22.6-58.6%), respectively. The results suggested that low dose ATG with low dose PTCy as GvHD prophylaxis in Haplo-PBSCT had promising activity. A prospective randomized trial is required to compare the efficacies of this regimen with ATG-based or PTCy-based regiments in Haplo-PBSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of hematologic malignancies (AML CR/blast cell≤20% high-risk MDS) were enrolled in this study. Diagnosis was according to the criteria of 2008 World Health Organization (WHO) classification of myeloid tumors.
2. Family members selected as donors were typed at the HLA-A, -B, -DQB1, -C and -DRB1 locus at high-resolution level. Haplotype was defined as recipient-donor number of HLA mismatches > 3.

3.14 to 70 years old. 4.Performance status scores no more than 2 (ECOG criteria). 5.Adequate organ function as defined by the following criteria: alanine transaminase （ALT）, aspartate transaminase（AST） and total serum bilirubin <2×ULN (upper limit of normal). Serum creatinine and blood urea nitrogen (BUN) <1.25×ULN.

6.Adequate cardiac function without acute myocardial infarction, arrhythmia or atrioventricular block, heart failure, active rheumatic heart disease and cardiac dilatation(the patients has been improved after treatment of the disease and are not expected to affect transplant can include in the study).

7.Absence of any other contraindications of stem cell transplantation. Willingness and ability to perform HSCT.

8.Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. DSA strong positive (titer >10000MFI)
2. Life expectancy < 3 months because of other severe diseases.
3. Presence of any fatal disease, including respiratory failure, heart failure, liver or kidney function failure.
4. Uncontrolled infection.
5. Pregnancy or breastfeeding.
6. Has enrolled in another clinical trials.
7. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2018-07-28 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
The cumulative incidences of acute GVHD | 100 days after transplantation
  The cumulative incidences of aGvHD was defined as the number and the ratio of the participants with aGVHD

SECONDARY OUTCOMES:
Leukocyte engraftment | 1 month
  Leukocyte engraftment:(was defined as the first of three consecutive days of peripheral white blood count >1000/ul.
Platelet engraftment | 1 month
  Platelet engraftment:(was defined as the first of seven consecutive days of platelet counts of >20000/ul.
Donor chimerism | 2 years
  Quantitative chimerism analyzes were performed using short-tandem-repeat-based polymerase chain reaction technique sat regular intervals for every 4 weeks after allografting in bone marrow.
Relapse incidence (RI) | 2 YEARS]
  RI was defined as the number and ratio of the participants with relapse after transplantation
chronic GVHD | 2 years
  cGvHD was diagnosed and graded according to the 2014 National Institutes of Health (NIH) consensus criteria: mild, moderate or severe respectively.The number and ratio of participants with cGVHD after transplatation
infection | 2 years
  CMV and EB infections(The number and ration of participants with infection after transplantaton)
OS | 2 years
  overall survival
DFS | 2 years
  disease free survival

CONTACTS AND LOCATIONS:
Overall Officials: xinpeng wang, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (6):
- China (6):
  - General Hospital of Jinan Military Command., Qinan, Shandong
  - Shanghai Ruijin Hospital, affiliated with the Medical School of Shanghai Jiaotong University,, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Xianmin Song, Shanghai, Shanghai Municipality
  - Shanghai Xinghua Hospital, affiliated with the Medical School of Shanghai Jiaotong University,, Shanghai, Shanghai Municipality
  - Shanghai tongji hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luznik L, Jalla S, Engstrom LW, Iannone R, Fuchs EJ. Durable engraftment of major histocompatibility complex-incompatible cells after nonmyeloablative conditioning with fludarabine, low-dose total body irradiation, and posttransplantation cyclophosphamide. Blood. 2001 Dec 1;98(12):3456-64. doi: 10.1182/blood.v98.12.3456. PMID 11719388
- [Background] Wang Y, Liu DH, Liu KY, Xu LP, Zhang XH, Han W, Chen H, Chen YH, Wang FR, Wang JZ, Sun YQ, Huang XJ. Long-term follow-up of haploidentical hematopoietic stem cell transplantation without in vitro T cell depletion for the treatment of leukemia: nine years of experience at a single center. Cancer. 2013 Mar 1;119(5):978-85. doi: 10.1002/cncr.27761. Epub 2012 Oct 23. PMID 23097265
- [Background] Wang Y, Chang YJ, Xu LP, Liu KY, Liu DH, Zhang XH, Chen H, Han W, Chen YH, Wang FR, Wang JZ, Chen Y, Yan CH, Huo MR, Li D, Huang XJ. Who is the best donor for a related HLA haplotype-mismatched transplant? Blood. 2014 Aug 7;124(6):843-50. doi: 10.1182/blood-2014-03-563130. Epub 2014 Jun 10. PMID 24916508
- [Background] Liu Q, Xuan L, Liu H, Huang F, Zhou H, Fan Z, Zhao K, Wu M, Xu L, Zhai X, Zhang F, Liu C, Sun J, Huang X. Molecular monitoring and stepwise preemptive therapy for Epstein-Barr virus viremia after allogeneic stem cell transplantation. Am J Hematol. 2013 Jul;88(7):550-5. doi: 10.1002/ajh.23452. Epub 2013 May 30. PMID 23564232
- [Background] Tischer J, Engel N, Fritsch S, Prevalsek D, Hubmann M, Schulz C, Zoellner AK, Bucklein V, Reibke R, Mumm F, Rieger CT, Hill W, Ledderose G, Stemmler HJ, Kohnke T, Jager G, Kolb HJ, Schmid C, Moosmann A, Hausmann A. Virus infection in HLA-haploidentical hematopoietic stem cell transplantation: incidence in the context of immune recovery in two different transplantation settings. Ann Hematol. 2015 Oct;94(10):1677-88. doi: 10.1007/s00277-015-2423-y. Epub 2015 Jun 10. PMID 26055139
- [Background] Luznik L, O'Donnell PV, Symons HJ, Chen AR, Leffell MS, Zahurak M, Gooley TA, Piantadosi S, Kaup M, Ambinder RF, Huff CA, Matsui W, Bolanos-Meade J, Borrello I, Powell JD, Harrington E, Warnock S, Flowers M, Brodsky RA, Sandmaier BM, Storb RF, Jones RJ, Fuchs EJ. HLA-haploidentical bone marrow transplantation for hematologic malignancies using nonmyeloablative conditioning and high-dose, posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2008 Jun;14(6):641-50. doi: 10.1016/j.bbmt.2008.03.005. PMID 18489989
- [Background] Ruggeri A, Labopin M, Bacigalupo A, Gulbas Z, Koc Y, Blaise D, Bruno B, Irrera G, Tischer J, Diez-Martin JL, Castagna L, Ciceri F, Mohty M, Nagler A. Bone marrow versus mobilized peripheral blood stem cells in haploidentical transplants using posttransplantation cyclophosphamide. Cancer. 2018 Apr 1;124(7):1428-1437. doi: 10.1002/cncr.31228. Epub 2018 Jan 23. PMID 29360162
- [Background] Bashey A, Zhang MJ, McCurdy SR, St Martin A, Argall T, Anasetti C, Ciurea SO, Fasan O, Gaballa S, Hamadani M, Munshi P, Al Malki MM, Nakamura R, O'Donnell PV, Perales MA, Raj K, Romee R, Rowley S, Rocha V, Salit RB, Solh M, Soiffer RJ, Fuchs EJ, Eapen M. Mobilized Peripheral Blood Stem Cells Versus Unstimulated Bone Marrow As a Graft Source for T-Cell-Replete Haploidentical Donor Transplantation Using Post-Transplant Cyclophosphamide. J Clin Oncol. 2017 Sep 10;35(26):3002-3009. doi: 10.1200/JCO.2017.72.8428. Epub 2017 Jun 23. PMID 28644773
- [Background] O'Donnell PV, Luznik L, Jones RJ, Vogelsang GB, Leffell MS, Phelps M, Rhubart P, Cowan K, Piantados S, Fuchs EJ. Nonmyeloablative bone marrow transplantation from partially HLA-mismatched related donors using posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2002;8(7):377-86. doi: 10.1053/bbmt.2002.v8.pm12171484.
- [Background] Brunstein CG, Gutman JA, Weisdorf DJ, Woolfrey AE, Defor TE, Gooley TA, Verneris MR, Appelbaum FR, Wagner JE, Delaney C. Allogeneic hematopoietic cell transplantation for hematologic malignancy: relative risks and benefits of double umbilical cord blood. Blood. 2010 Nov 25;116(22):4693-9. doi: 10.1182/blood-2010-05-285304. Epub 2010 Aug 4. PMID 20686119
- [Background] Chen J, Wang RX, Chen F, Sun AN, Qiu HY, Jin ZM, Tang XW, Han Y, Fu ZZ, He GS, Miao M, Ma X, Wu DP. Combination of a haploidentical SCT with an unrelated cord blood unit: a single-arm prospective study. Bone Marrow Transplant. 2014 Feb;49(2):206-11. doi: 10.1038/bmt.2013.154. Epub 2013 Oct 21. PMID 24141650
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Martin PJ, Lee SJ, Przepiorka D, Horowitz MM, Koreth J, Vogelsang GB, Walker I, Carpenter PA, Griffith LM, Akpek G, Mohty M, Wolff D, Pavletic SZ, Cutler CS. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: VI. The 2014 Clinical Trial Design Working Group Report. Biol Blood Marrow Transplant. 2015 Aug;21(8):1343-59. doi: 10.1016/j.bbmt.2015.05.004. Epub 2015 May 15. PMID 25985921